CLINICAL TRIAL: NCT00755833
Title: A Prospective, Multicentre, Open Label, Un-controlled , Observational, 12-month Study in Subjects Using: NovoMix® 50 (Biphasic Insulin Aspart 50) for Treatment of Type 2 Diabetes Mellitus in Slovenia
Brief Title: Observational Study of NovoMix® 50 for Treatment of Type 2 Diabetics for 12 Months
Status: Completed | Type: Observational
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Other Study IDs: BIASP-3674
Record Dates: First submitted 2008-09-18; First posted 2008-09-19 (Estimated); Last update posted 2016-10-31 (Estimated); Status verified 2016-10

CONDITIONS: Diabetes; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- A
  Interventions: Drug: biphasic insulin aspart 50

INTERVENTIONS:
Drug: biphasic insulin aspart 50 — Efficacy and safety data collection in connection with the use of the drug NovoMix® 50 in daily clinical practice.
  Other Names: NovoMix® 50

SUMMARY:
This study is conducted in Europe. The aim of this observational study is to evaluate the blood glucose control when using NovoMix® 50 up to 12 months after initiation subjects with type 2 diabetes currently on a therapy with human biphasic insulin. An additional objective is also to observe the different regimes of starting and maintaining the treatment with NovoMix® 50 during one year.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes treated with biphasic human insulin with or without metformin
* Inadequate glycaemic control or is experiencing hypoglycaemic events or would, in the physician's opinion, benefit from treatment with NovoMix® 50

Exclusion Criteria:

* Subjects with diagnosed type 1 diabetes mellitus
* Subjects treated with short acting or intermediate acting human insulin or any insulin analogue
* Subjects who are unlikely to comply with study description, e.g. uncooperative attitude, inability to come for regular visits
* Subjects with a hypersensitivity to biphasic insulin aspart 50 (NovoMix® 50 )or to any of the excipients
* Women of childbearing potential, who are pregnant, breast-feeding or intend to become pregnant within next 12 months

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Type 2 diabetes patients from both general and speciality practice settings who have been deemed appropriate to receive NovoMix® 50 as new treatment and as part of routine out-patient care by the prescribing physician.
Sampling Method: Non-Probability Sample
Enrollment: 270 (Actual)
Dates: Start 2008-09; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
Change in HbA1c | At 0, 3, 6, 9, 12 months

SECONDARY OUTCOMES:
Percentage of subjects achieving target HbA1c | At 0, 3, 6, 9, 12 months
Change in FPG (fasting plasma glucose) | At 0, 3, 6, 9, 12 months
Change in PPG (postprandial glucose) | At 0, 3, 6, 9, 12 months
Change in number of hypoglycaemic events | At 0, 3, 6, 9, 12 months
Change in insulin presentation | At 0, 3, 6, 9, 12 months
Dose and number of injections | At 0, 3, 6, 9, 12 months
Number of ADRs (adverse drug reaction) | At 0, 3, 6, 9, 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (1):
- Novo Nordisk Investigational Site, Ljubljana, Slovenia

REFERENCES:
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com